CLINICAL TRIAL: NCT00362765
Title: Assessment of Insulin Sensitivity in Type 2 Diabetics Treated With Metformin, Fenofibrate and Their Combination.
Brief Title: Fenofibrate and Metformin Insulin Sensitivity in Type 2 Diabetics Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was prematurely terminated, due to difficulties in the recruitment of T2DM patients who are not under statin therapy at inclusion.
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Philippe Jais, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C LF23-0121 05 03; 2005-003347-31
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Type 2 Diabetes; Dyslipidemia
Keywords: Type 2 Diabetes; Dyslipidemia; Hyperinsulinemic; Clamp; Metformin; Fenofibrate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Fenofibrate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate; Drug: Metformin
- 2 (Active Comparator)
  Interventions: Drug: Fenofibrate
- 3 (Active Comparator)
  Interventions: Drug: Metformin
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate — 160 mg
  Arms: 1; 2
Drug: Metformin — 2000 mg
  Arms: 1; 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
Double-blind, randomized placebo-controlled study in type 2 diabetes and dyslipidemic patients.Patients will be randomized to one of four treatment arms for 16 weeks: placebo, fenofibrate, metformin, or metformin and fenofibrate combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus and dyslipidemia.

Exclusion Criteria:

* Type 1 diabetes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Endogenous Glucose Production (EGP) and Glucose Disposal Rate (GDR) by two-step hyperinsulinemic euglycemic clamp (HEC) | 16 weeks

SECONDARY OUTCOMES:
Gluconeogenesis, Glycogenolysis, Skeletal muscle and liver fat content, Abdominal fat content, Body energy expenditure and respiratory quotient, Lipids and glycemic parameters | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (3):
- Site 2, Turku, Finland
- Site 3, Dublin, Ireland
- Site 1, Pisa, Italy